CLINICAL TRIAL: NCT05396079
Title: Effect of Tahini Consumption on Oxidative Stress and Inflammation Markers as Well as Endothelial Function and Arterial Stiffness in Patients With Type 2 Diabetes
Brief Title: Effect of Tahini in Oxidative Stress and Endothelial Function in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, PANAGIOTIS KANELLOS, Postdoctoral Researcher, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-03

CONDITIONS: Oxidative Stress; Endothelial Function; Blood Pressure; Arterial Stiffness; Blood Glucose; Diabetes Mellitus, Type 2
Keywords: tahini; sesame; antioxidants; postprandial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; SeSAME syndrome | interventions — Bread; Margarine; Cheese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tahini and bread (Experimental): After an overnight fast (10-12 h), participants will come tο the lab and, after a 10-min resting period in the supine position in a quiet room with temperature a constant 20-25 °C, assessment of blood pressure, pulse rate, hemodynamic parameters, and endothelial function will be performed.
  Then, an intravenous cannula will be inserted into a forearm vein and a baseline blood sample will be collected (time 0) as well as urine sample will be also collected. Afterward, each patient will consume 2 slices of white bread with 50 g of tahini and collection of the blood and urine sample will be repeated 1,2, 3 and 4 h postprandially. Assessment of blood pressure, pulse rate, hemodynamic parameters, and endothelial function will be also repeated at the end of the trial. During the trial, patients will not be allowed to eat or drink anything apart from water.
  Interventions: Other: tahini and bread
- Margarine, cheese and bread (Experimental): After an overnight fast (10-12 h), participants will come tο the lab and, after a 10-min resting period in the supine position in a quiet room with temperature a constant 20-25 °C, assessment of blood pressure, pulse rate, hemodynamic parameters, and endothelial function will be performed.
  Then, an intravenous cannula will be inserted into a forearm vein and a baseline blood sample will be collected (time 0) as well as urine sample will be also collected. Afterward, each patient will consume 2 slices of white bread with 46 g of margarine and 38 g of lowfat cheese and collection of the blood and urine sample will be repeated 1,2, 3 and 4 h postprandially. Assessment of blood pressure, pulse rate, hemodynamic parameters, and endothelial function will be also repeated at the end of the trial. During the trial, patients will not be allowed to eat or drink anything apart from water.
  Interventions: Other: margarine, cheese and bread

INTERVENTIONS:
Other: tahini and bread — Fifthy grams of tahini with 2 slices of white bread
  Arms: Tahini and bread
Other: margarine, cheese and bread — 46 g of margarine and 38 g of cheese with 2 slices of white bread
  Arms: Margarine, cheese and bread

SUMMARY:
Cardiovascular disease (CVD), a cluster of disorders that affect heart and blood vessels, is the leading cause of morbidity and mortality around the world and is responsible for 17.9 million deaths annually worldwide. CVD risk factors can be modifiable (nutrition, physical activity, obesity, smoking, hyperlipidemia, hypertension and diabetes) and non-modifiable (age, gender, ethnicity, family history and socioeconomic status). Chronic exposure to CVD risk factors induces oxidative stress and promotes inflammation. In addition, endothelial cells in response to the inflammatory reaction secrete growth factors, leading to the destruction of vascular endothelium and promoting atherogenesis.

Oxidative stress refers to the imbalance between anti-oxidant and pro-oxidant compounds, with predominance of the pro-oxidant ones. Reactive Oxygen Species overproduction has been implicated in pathogenesis and complications of numerous diseases including diabetes, cardiovascular diseases, cancer, neurodegenerative diseases and chronic kidney disease.

Moreover, endothelium consists of a single layer of endothelial cells; it is the natural barrier between blood and tissues and also an endocrine organ. It plays a key role in vascular homeostasis by maintaining a balance between vasodilation and vasoconstriction and is responsible for fluid filtration, blood vessel tone, hormone trafficking, hemostasis, regulation of blood flow and growth of blood vessels. Thus, reductions in endothelial function are detrimental and predict and precede the development of overt CVD.

Sesame belongs to Pedaliaceae family and can be consumed in different forms such as seeds, oil or tahini, i.e., a 100 % peeled, ground and roasted sesame paste. Tahini is rich in polyunsaturated fatty acids, proteins, vitamin E and lignans, such as sesamin, sesamolin and sesamol. Recent studies have indicated that tahini consumption can lower blood pressure and pulse rate and improve endothelial function and glycemic response in healthy males postprandially.

However, only two studies are available in the current literature concerning the effect on diabetes, one of them in patients with type 2 diabetes and one in diabetic animal model. Thus, the aim of the present study is to investigate the effect of tahini consumption on oxidative stress, blood pressure, endothelial function and arterial stiffness in patients with type 2 diabetes postprandially.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), a cluster of disorders that affect heart and blood vessels, is the leading cause of morbidity and mortality around the world and is responsible for 17.9 million deaths annually worldwide. CVD includes coronary heart disease, peripheral arterial disease, cerebrovascular disease, rheumatic heart disease, congenital heart disease, deep vein thrombosis and pulmonary embolism. CVD risk factors can be modifiable (nutrition, physical activity, obesity, smoking, hyperlipidemia, hypertension and diabetes) and non-modifiable (age, gender, ethnicity, family history and socioeconomic status). Chronic exposure to CVD risk factors induces oxidative stress and promotes inflammation. In addition, endothelial cells in response to the inflammatory reaction secrete growth factors, leading to the destruction of vascular endothelium and promoting atherogenesis.

Oxidative stress refers to the imbalance between anti-oxidant and pro-oxidant compounds, with predominance of the pro-oxidant ones. These compounds are also called Reactive Oxygen Species (ROS) or free radicals and are unstable atoms or molecules. Their generation, as products of normal cellular metabolism, occurs naturally by endogenous sources (e.g. mitochondria, peroxisomes and endoplasmic reticulum) through enzymatic and non-enzymatic reactions. Furthermore, exogenous sources implicated in free radical production are air pollution, alcohol consumption, tobacco smoking, ultraviolet light exposure, industrial solvents and others. Free radical production is regulated by the well-organized human endogenous enzymatic and non-enzymatic antioxidant system, along with the exogenous antioxidants found in food. However, in some cases antioxidant system fails to eliminate ROS overproduction and can consequently induce serious damage to important for life biomolecules (DNA, lipids, proteins), leading to cell injury and death. Thus, ROS overproduction has been implicated in pathogenesis and complications of numerous diseases including diabetes, cardiovascular diseases, cancer, neurodegenerative diseases and chronic kidney disease.

Moreover, endothelium consists of a single layer of endothelial cells; it is the natural barrier between blood and tissues and also an endocrine organ. It plays a key role in vascular homeostasis by maintaining a balance between vasodilation and vasoconstriction. Moreover, vascular endothelium is responsible for fluid filtration, blood vessel tone, hormone trafficking, hemostasis, regulation of blood flow and growth of blood vessels. Thus, reductions in endothelial function are detrimental and predict and precede the development of overt CVD.

Sesame belongs to Pedaliaceae family and can be consumed in different forms such as seeds, oil or tahini, i.e., a 100 % peeled, ground and roasted sesame paste. Sesame seeds are rich in polyunsaturated fatty acids (PUFAs), proteins, vitamin E and lignans, such as sesamin, sesamolin and sesamol. Recent studies have highlighted the antioxidant, antihypertensive, hypolipidemic and appetite control properties of sesame seeds and sesame oil. Moreover, few studies have investigated the effect of sesame consumption on blood pressure, endothelial function and arterial stiffness in human population. According to a metanalysis, sesame consumed in form of seed, oil, capsule or bar decreased both systolic blood pressure (SBP) and diastolic blood pressure (DBP), while sesame oil consumption was found to improve endothelial function both in the postprandial state and after long term consumption in hypertensive men.

Regarding the consumption of tahini and its effect on human health, only a few studies are available in the current literature. The most recent of them have indicated that tahini consumption can lower blood pressure and pulse rate and improve endothelial function and glycemic response in healthy males postprandially. However, only two studies are available in the current literature concerning the effect on diabetes, one of them in patients with type 2 diabetes and one in diabetic animal model. Thus, the aim of the present study is to investigate the effect of tahini consumption on oxidative stress, blood pressure, endothelial function and arterial stiffness in patients with type 2 diabetes postprandially.

ELIGIBILITY:
Inclusion Criteria:

* minimum period from diagnosis three years
* good glycemic control (HbA1c <7%)
* taking a stable anti-diabetic treatment for the last 3 months (anti-diabetic tablets only)

Exclusion Criteria:

-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Concentration of urinary 8-iso-prostaglandin F2a | Four hours after consumption of both meals
  We will measure the concentration of urinary 8-iso-prostaglandin F2a by using Elisa kit
Assessment of Flow-Mediated Dilatation | Four hours after consumption of both meals
  We will assess the FMD by high-resolution ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: NIKOLAOS K TENTOLOURIS, PROF, Study Director — Diabetes Center, Medical School, National and Kapodistrian University of Athens
Locations (1):
- Panagiotis Kanellos, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sies H. Oxidative stress: a concept in redox biology and medicine. Redox Biol. 2015;4:180-3. doi: 10.1016/j.redox.2015.01.002. Epub 2015 Jan 3. PMID 25588755
- [Background] Kumar, S., & Pandey, A. (2015). Free Radicals: Health Implications and their Mitigation by Herbals. British Journal Of Medicine And Medical Research, 7(6), 438-457. doi: 10.9734/bjmmr/2015/16284
- [Background] Phaniendra A, Jestadi DB, Periyasamy L. Free radicals: properties, sources, targets, and their implication in various diseases. Indian J Clin Biochem. 2015 Jan;30(1):11-26. doi: 10.1007/s12291-014-0446-0. Epub 2014 Jul 15. PMID 25646037
- [Background] Birben E, Sahiner UM, Sackesen C, Erzurum S, Kalayci O. Oxidative stress and antioxidant defense. World Allergy Organ J. 2012 Jan;5(1):9-19. doi: 10.1097/WOX.0b013e3182439613. Epub 2012 Jan 13. PMID 23268465
- [Background] Willcox JK, Ash SL, Catignani GL. Antioxidants and prevention of chronic disease. Crit Rev Food Sci Nutr. 2004;44(4):275-95. doi: 10.1080/10408690490468489. PMID 15462130
- [Background] Ravarotto V, Simioni F, Pagnin E, Davis PA, Calo LA. Oxidative stress - chronic kidney disease - cardiovascular disease: A vicious circle. Life Sci. 2018 Oct 1;210:125-131. doi: 10.1016/j.lfs.2018.08.067. Epub 2018 Aug 31. PMID 30172705
- [Background] Zoumpoulakis, P., Sinanoglou, V., Batrinou, A., Strati, I., Miniadis-Meimaroglou, S., & Sflomos, K. (2012). A combined methodology to detect γ-irradiated white sesame seeds and evaluate the effects on fat content, physicochemical properties and protein allergenicity. Food Chemistry, 131(2), 713-721. doi: 10.1016/j.foodchem.2011.09.049
- [Background] Namiki M. Nutraceutical functions of sesame: a review. Crit Rev Food Sci Nutr. 2007;47(7):651-73. doi: 10.1080/10408390600919114. PMID 17943496
- [Background] Raeisi-Dehkordi, H., Mohammadi, M., Moghtaderi, F., & Salehi-Abargouei, A. (2018). Do sesame seed and its products affect body weight and composition? A systematic review and meta-analysis of controlled clinical trials. Journal Of Functional Foods, 49, 324-332. doi: 10.1016/j.jff.2018.08.036
- [Background] Pathak N, Rai AK, Kumari R, Bhat KV. Value addition in sesame: A perspective on bioactive components for enhancing utility and profitability. Pharmacogn Rev. 2014 Jul;8(16):147-55. doi: 10.4103/0973-7847.134249. PMID 25125886
- [Background] Gouveia Lde A, Cardoso CA, de Oliveira GM, Rosa G, Moreira AS. Effects of the Intake of Sesame Seeds (Sesamum indicum L.) and Derivatives on Oxidative Stress: A Systematic Review. J Med Food. 2016 Apr;19(4):337-45. doi: 10.1089/jmf.2015.0075. PMID 27074618
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Park KH, Park WJ. Endothelial Dysfunction: Clinical Implications in Cardiovascular Disease and Therapeutic Approaches. J Korean Med Sci. 2015 Sep;30(9):1213-25. doi: 10.3346/jkms.2015.30.9.1213. Epub 2015 Aug 13. PMID 26339159
- [Background] Kruger-Genge A, Blocki A, Franke RP, Jung F. Vascular Endothelial Cell Biology: An Update. Int J Mol Sci. 2019 Sep 7;20(18):4411. doi: 10.3390/ijms20184411. PMID 31500313
- [Background] Rajendran P, Rengarajan T, Thangavel J, Nishigaki Y, Sakthisekaran D, Sethi G, Nishigaki I. The vascular endothelium and human diseases. Int J Biol Sci. 2013 Nov 9;9(10):1057-69. doi: 10.7150/ijbs.7502. eCollection 2013. PMID 24250251
- [Background] Alipoor B, Haghighian MK, Sadat BE, Asghari M. Effect of sesame seed on lipid profile and redox status in hyperlipidemic patients. Int J Food Sci Nutr. 2012 Sep;63(6):674-8. doi: 10.3109/09637486.2011.652077. Epub 2012 Jan 23. PMID 22263599
- [Background] Khosravi-Boroujeni H, Nikbakht E, Natanelov E, Khalesi S. Can sesame consumption improve blood pressure? A systematic review and meta-analysis of controlled trials. J Sci Food Agric. 2017 Aug;97(10):3087-3094. doi: 10.1002/jsfa.8361. Epub 2017 May 12. PMID 28387047
- [Background] Kamal-Eldin A, Frank J, Razdan A, Tengblad S, Basu S, Vessby B. Effects of dietary phenolic compounds on tocopherol, cholesterol, and fatty acids in rats. Lipids. 2000 Apr;35(4):427-35. doi: 10.1007/s11745-000-541-y. PMID 10858028
- [Background] Wu WH, Kang YP, Wang NH, Jou HJ, Wang TA. Sesame ingestion affects sex hormones, antioxidant status, and blood lipids in postmenopausal women. J Nutr. 2006 May;136(5):1270-5. doi: 10.1093/jn/136.5.1270. PMID 16614415
- [Background] Khalesi S, Paukste E, Nikbakht E, Khosravi-Boroujeni H. Sesame fractions and lipid profiles: a systematic review and meta-analysis of controlled trials. Br J Nutr. 2016 Mar 14;115(5):764-73. doi: 10.1017/S0007114515005012. Epub 2016 Jan 13. PMID 26758593
- [Background] Hirata F, Fujita K, Ishikura Y, Hosoda K, Ishikawa T, Nakamura H. Hypocholesterolemic effect of sesame lignan in humans. Atherosclerosis. 1996 Apr 26;122(1):135-36. doi: 10.1016/0021-9150(95)05769-2. No abstract available. PMID 8724120
- [Background] Neves Ribeiro D, Goncalves Alfenas Rde C, Bressan J, Brunoro Costa NM. The effect of oilseed consumption on appetite and on the risk of developing type 2 diabetes mellitus. Nutr Hosp. 2013 Mar-Apr;28(2):296-305. doi: 10.3305/nh.2013.28.2.6309. PMID 23822678
- [Background] Karatzi K, Stamatelopoulos K, Lykka M, Mantzouratou P, Skalidi S, Zakopoulos N, Papamichael C, Sidossis LS. Sesame oil consumption exerts a beneficial effect on endothelial function in hypertensive men. Eur J Prev Cardiol. 2013 Apr;20(2):202-8. doi: 10.1177/2047487312437625. Epub 2012 Jan 25. PMID 22345690
- [Background] Sakketou EI, Baxevanis GK, Tentolouris NK, Konstantonis GD, Karathanos VT, Fragkiadakis GA, Kanellos PT. Tahini consumption affects blood pressure and endothelial function in healthy males. J Hum Hypertens. 2022 Dec;36(12):1128-1132. doi: 10.1038/s41371-021-00624-2. Epub 2021 Oct 27. PMID 34707227
- [Background] Baxevanis, G.K., Sakketou, EK.I., Tentolouris, N.K. et al. Tahini consumption improves metabolic and antioxidant status biomarkers in the postprandial state in healthy males. Eur Food Res Technol 247, 2721-2728 (2021). https://doi.org/10.1007/s00217-021-03828-5